CLINICAL TRIAL: NCT04816604
Title: An Open-label Extension Study Evaluating the Long-term Safety and Efficacy of Oral Inhalation of GB002 for the Treatment of WHO Group 1 Pulmonary Arterial Hypertension (PAH)
Brief Title: Open-label Extension Study of GB002 in Adult Subjects With Pulmonary Arterial Hypertension (PAH)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GB002, Inc., a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB002-2102
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: seralutinib
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- GB002 (seralutinib) (Experimental): GB002 (seralutinib) inhaled orally twice per day (BID)
  Interventions: Drug: GB002 (seralutinib); Device: Generic Dry Powder Inhaler

INTERVENTIONS:
Drug: GB002 (seralutinib) — Capsule containing GB002 (seralutinib)
Device: Generic Dry Powder Inhaler — Generic dry powder inhaler for GB002 (seralutinib) delivery

SUMMARY:
This open-label extension study will evaluate the long-term effects of GB002 (seralutinib) in subjects who previously participated in a GB002 PAH study.

ELIGIBILITY:
Inclusion Criteria:

Type of Subject and Disease Characteristics

1. Subjects must have completed a prior GB002 PAH study and, in the opinion of the Investigator and Sponsor, have been compliant with study procedures and have completed treatment with IP through parent study end-of-treatment (EOT) visit.
2. Treatment with standard of care PAH disease-specific background therapies (stable dose).

   Informed Consent
3. Review and signature of an IRB-approved informed consent form.

Exclusion Criteria:

Medical Conditions

1. Persistent and clinically significant systemic hypertension or hypotension.
2. Interval history of newly developed left-sided heart disease.
3. Potentially life-threatening cardiac arrhythmia with an ongoing risk.
4. Uncontrolled bacterial, viral, or fungal infections which require systemic therapy.
5. Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or GB002 administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
6. History of portopulmonary hypertension or portal hypertension due to cirrhosis classified as Child-Pugh Class A or higher.
7. Subjects with a history of severe milk protein allergy. In addition, subjects with known intolerance or hypersensitivity to lactose who, in the opinion of the investigator, may experience severe symptoms following the ingestion of lactose.
8. Current use of inhaled tobacco and/or inhaled marijuana. Ingestible or topical marijuana is allowed, per local restrictions and regulations.
9. Current alcohol use disorder as defined by DSM-5, and/or history of current utilization of drugs of abuse (amphetamines, methamphetamines, cocaine, phencyclidine [PCP]).
10. Have any other condition or reason that, in the opinion of the Investigator and/or the Sponsor's Medical Monitor (or designee), would prohibit the subject from participating in the study.

    Diagnostic Assessments
11. Chronic renal insufficiency
12. Hemoglobin (Hgb) concentration <8.5 g/dL.
13. Absolute neutrophil count (ANC) < 1x 10^9/L.
14. Platelet count <50 x 10^9/L.

    Prior Therapy
15. Use of inhaled prostanoids.
16. Chronic use of oral anticoagulants (ie, vitamin K antagonist such as warfarin or novel oral anticoagulant [NOAC]/direct oral anticoagulant [DOAC]).
17. Chronic use of any prohibited medication.

NOTE: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events | From first dose of study drug up to 80 months or availability of commercial product

SECONDARY OUTCOMES:
Change from Baseline Over Time on the Six-Minute Walk Test (6MWT) | Baseline, up to 80 months or availability of commercial product
  Change in the distance achieved on the 6MWT (Δ6MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aranda, Study Director — Gossamer Bio Inc.
Locations (28):
- United States (15):
  - University of California, Davis Medical Center, Sacramento, California
  - Medical Corporation, Santa Barbara, California
  - Mayo Clinic, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Inc., Oklahoma City, Oklahoma
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
- Australia (2):
  - Royal Hobart Hospital, Hobart, Tasmania
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
- Všeobecná fakultní nemocnice v Praze, Prague, Czechia
- AP-HP Hôpital de Bicêtre, Le Kremlin-Bicêtre, France
- Germany (5):
  - DRK Kliniken Berlin, Berlin
  - Universitaetsklinikum Giessen und Marburg GmbH - Medizinische Klinik IV und V, Giessen
  - Klinik für Pneumologie, Klinisches Studienzentrum Medizinische Hochschule, Hanover
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Klinik und Poliklinik f. Innere Medizin II Universitätsklinikum Regensburg, Regensburg
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Imperial College Healthcare NHS Trust - Hammersmith Medicines Research Limited, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sitbon O, Sahay S, Escribano Subias P, Zolty RL, Kingrey JF, Ryan JJ, Sobol I, Sood N, Benza RL, Channick RN, Chin KM, Frantz RP, Ghofrani HA, Hemnes AR, McLaughlin VV, Vachiery JL, Zamanian RT, Ter Veer A, Roscigno RF, Mottola D, Parsley E, Aranda R, Zisman LS, Howard LS; TORREY Study Investigators. Seralutinib for the Treatment of Pulmonary Arterial Hypertension in Adults: TORREY Open-Label Extension Study. Adv Ther. 2025 Oct;42(10):5104-5123. doi: 10.1007/s12325-025-03297-2. Epub 2025 Aug 11. PMID 40788460